CLINICAL TRIAL: NCT06703931
Title: Evaluation of PERThermodiag® Medical Device for CT Temperature Measurement and Anomaly Detection Compared to Reference Methods in Critical Care Hospitalized Patients: a Comparative, Multi-center Interventional Study
Brief Title: Performance Study of the Thermodiag Solution for Body Temperature Measurement
Acronym: ThermodiagPERF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: F2D Medical (Industry)
Collaborators: Clinact Multihealth (Unknown); Digital Medical Hub (Other)
Responsible Party: Principal Investigator, Daniel DA SILVA, Principal Investigator, Delafontaine Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A02014-41_NIFC
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Temperature Change, Body; Emergency Department Visit
Keywords: Temperature; Body temperature; Monitoring temperature; multisensors; Actimetry; Actigraphy; Heart rate; Continuous measurement; Contextualized measure; Dedicated machine learning model; Machine Learning
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, multi-centre interventional clinical investigation
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temperature Monitor (Experimental): Patients included in the study will have their temperature measured simultaneously during their stay in intensive care, with Thermodiag(R) and with the reference medical device.
  Interventions: Device: Measures performed on all subjects

INTERVENTIONS:
Device: Measures performed on all subjects — In intensive care Medics will use a reference medical device and Thermodiag®. Simultaneous and synchronised measurements will be taken every minute.

SUMMARY:
The goal of this prospective, comparative, multi-centre interventional clinical investigation, is to evaluate the performance of the Thermodiag® medical device, compared with reference methods, for continuous measurement of core temperature in critical care patients. The main question it aims to answer is to develop non-invasive alternatives to the current methods of measuring core body, to reduce health risks, and overcome various other limitations (as infection, bleeding, thrombosis and local reactions).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years;
* Female or male patients;
* Patients hospitalised in a critical care unit as defined by the Public Health Code of the Republic of France, Article R6123-33: 'The critical care activity consists of the care of patients who present or are likely to present one or more acute failures directly threatening the vital or functional prognosis and which may require recourse to one or more methods of substitution'.
* Patients affiliated to the social security system or beneficiaries of such a system, where applicable, in accordance with local regulations;
* Voluntary patients - or trusted person/family member/relative who have given oral and written consent after being informed by the investigator of the research.

Exclusion Criteria:

* Patients with a corpulence or physical characteristics responsible for a 'tourniquet' effect: arm circumference greater than 47 centimetres;
* Patients with burns on the arm (location for Thermodiag® measurement);
* Patients with particularly sensitive or affected skin in the biceps or armpit (left and right);
* Patients undergoing an MRI examination;
* Patients undergoing extracorporeal circulation;
* Patients with a history of allergy to silicone;
* Patients with active implantable medical devices such as pacemakers, defibrillators, etc. ;
* Patients undergoing dialysis;
* Patients with a tattoo in the area where the investigational device will be worn (arm);
* Patients currently excluded from another protocol or taking part in another interventional research study;
* Pregnant or breast-feeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-26 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Body temperature Measurement | Every minute from the enrollment to the end of medical treatment (estimated time : 8 days)
  The degree of agreement between the two medical devices (Thermodiag® versus reference method in the hospital unit) will be assessed (expected measure is less than 0.1°C).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier De Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier Intercommunal - Nord-Ardennes, Charleville-Mézières
  - Hôpital Privé de l'Ouest Parisien, Trappes
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: No
According to GDPR Regulation 2016, patients data are sensitive. Sponsor is requirred to return them to facilities or to destroy them. That's why no patients data are planed to be shared.